CLINICAL TRIAL: NCT02032628
Title: DNA Methylation and Cancer Prevention: Duration and Intensity of Exercise
Acronym: GEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Angela Bryan, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PQA-5; 1R01CA179963-01 (NIH)
Record Dates: First submitted 2013-12-16; First posted 2014-01-10 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: DNA Methylation
Keywords: epigenetics; cancer; exercise; intensity; duration
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Intensity/Longer Duration (Experimental): Exercise at higher intensity (~75% of VO2max) for 40 minute bouts 4 times per week
  Interventions: Behavioral: Exercise
- High Intensity/Lower Duration (Experimental): Exercise at high intensity (~75% of VO2max) for 20 minute bouts 4 times per week
  Interventions: Behavioral: Exercise
- Lower Intensity/Higher Duration (Experimental): Exercise at lower intensity (~55% of VO2max) for 40 minute bouts 4 times per week
  Interventions: Behavioral: Exercise
- Low Intensity/Low Duration (Experimental): Exercise at lower intensity (~55% of VO2max) for 20 minute bouts 4 times per week
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The investigators will measure changes in DNA methylation as a result of four different intervention groups, i.e, high/longer, low/longer, high/shorter, low/shorter.
  Other Names: GEM

SUMMARY:
Specific aim 1. Using a fully crossed 2 (intensity) X 2 (duration) design, the investigators will demonstrate a dose-response relationship between volume of aerobic exercise and changes in DNA methylation over four months among previously sedentary women.

Specific aim 2. There are no published data on the extent to which positive effects of exercise on methylation might decay if exercise is not continued. The investigators will gather data on the natural history of methylation decay after training.

DETAILED DESCRIPTION:
Specific aim 1. Using a fully crossed 2 (intensity) X 2 (duration) design, the investigators will demonstrate a dose-response relationship between volume of aerobic exercise and changes in DNA methylation over four months among previously sedentary women.

* Hypothesis 1: The investigators predict that there will be an interaction between intensity and duration characterized by a dose-dependent response to total exercise volume, such that women will experience the greatest improvements in methylation at high intensity/high duration (16.4 kcal/kg/week) and the least improvements in methylation at low intensity/low duration (5.6 kcal/kg/week).
* Hypothesis 2: The investigators predict that there will be a main effect of exercise duration, such that women exercising for 40 minutes/session, 4 sessions per week will show more improvement in DNA methylation compared with women exercising for 20 minutes/session, 4 sessions per week.
* Hypothesis 3: The investigators predict that there will be a main effect of exercise intensity, such that women exercising at 75% of VO2max will show more improvement in DNA methylation compared with women exercising at 55% of VO2max.

Specific aim 2. There are no published data on the extent to which positive effects of exercise on methylation might decay if exercise is not continued. The investigators will gather data on the natural history of methylation decay after training.

• Hypothesis 4: At six months following the end of supervised exercise, the investigators will assess the influence of the different levels of initial training and the passage of time on DNA methylation, covarying whether or not participants continued to exercise. It is predicted that the highest volume group will show the greatest persistence of positive changes in DNA methylation. Alternatively, it is possible that all four groups will return to baseline methylation levels of methylation, and there will be no difference in methylation at 6 months following the end of supervised exercise.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 30-45
* Sedentary (i.e., < 40 minutes per week of moderate physical activity in the past 6-months; this criterion will be relaxed to <60 minutes per week if it limits enrollment)
* Menstruating regularly (not amenorrheic or dysmenorrheic)
* Non-smokers
* Willing to accept random assignment to condition
* Willing to provide blood and saliva samples for epigenetic analysis
* Willing to and physically capable of safely engaging in moderate exercise activity (i.e., no injuries, physical impairments, or pre-existing contraindications) as assessed by a study physician
* Able to successfully complete a VO2max test without evidence of cardiac or other abnormalities
* Planning to remain in the Denver metro area for the next 10 months

Exclusion Criteria:

* Have a BMI > 35kg/m2
* Are diabetic or on a restricted diet
* Have uncontrolled hypertension defined as resting systolic BP >150 mmHg or diastolic BP>90 mmHg (to be assessed during physical exam, not on phone screen). (Participants who do not meet these criteria at first screening will be re-evaluated, including after follow-up evaluation by the primary care physician with initiation or adjustment of anti-hypertensive medications)
* Have a cardiovascular or respiratory disease including subjective or objective indicators of ischemic heart disease (e.g., angina, ST segment depression) or serious arrhythmias at rest or during the maximal exercise test (VO2max). (Participants who do not meet these criteria at first screening will be re-evaluated; follow-up evaluation must include diagnostic testing (e.g., thallium stress test) with interpretation by a cardiologist)
* Have a history of breast neoplasia
* Are currently receiving treatment for any type of cancer
* Are on psychotropic medications
* Are currently under treatment for any psychiatric disorder
* Are currently under treatment for alcohol or drug abuse
* Are currently pregnant or attempting to become pregnant in the next 6-months

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2014-01; Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
DNA METHYLATION | 4 months post-exercise initiation and 6 months after the end of the exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bryan, PhD, Principal Investigator — University of Colorado, Boulder; Wendy kohrt, PhD, Principal Investigator — UColoradoDenver
Locations (1):
- Image Lab/ University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Gillman AS, Stevens CJ, Bryan AD. Women's exercise identity increases after a 16-week exercise RCT and is linked to behavior maintenance at follow-up. Psychol Sport Exerc. 2021 May;54:101888. doi: 10.1016/j.psychsport.2021.101888. Epub 2021 Jan 12. PMID 33633498
- [Derived] Stevens CJ, Gillman AS, Giordano GR, Bryan AD. Modeling longitudinal variation in affective response to exercise across a 16-week randomized control trial (RCT). Health Psychol. 2021 Dec;40(12):928-939. doi: 10.1037/hea0001023. Epub 2020 Sep 24. PMID 32969699